CLINICAL TRIAL: NCT04672928
Title: A Clinical Study to Evaluate the Efficacy and Safety of IBI318 in Combination With Paclitaxel Versus Placebo in Combination With Paclitaxel in Patients With Small Cell Lung Cancer Who Have Failed First-line or Above Chemotherapies
Brief Title: A Phase Ib/III Clinical Study to Evaluate the Efficacy and Safety of IBI318 in Combination With Paclitaxel Versus Placebo in Combination With Paclitaxel in Patients With Small Cell Lung Cancer Who Have Failed First-line or Above Chemotherapies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI318C302
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI318 in combination with paclitaxel (Experimental)
  Interventions: Drug: paclitaxel; Drug: IBI318

INTERVENTIONS:
Drug: paclitaxel — 80mg/m^2,iv,Q4W
Drug: IBI318 — 300mg,iv,Q4W

SUMMARY:
This study is a phase Ib/III clinical study to evaluate the efficacy and safety of recombinant fully human anti-programmed cell death receptor 1 (PD-1) and anti-programmed cell death ligand 1 (PD-L1) bispecific antibody injection (IBI318) in combination with paclitaxel versus placebo in combination with paclitaxel in subjects with small cell lung cancer who have failed first-line or above chemotherapies.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the Informed Consent Form;
2. Male or female ≥ 18 and≤75 years of age;
3. Life expectancy ≥ 12 weeks;
4. Pathologically confirmed limited or extensive stage small cell lung cancer according to Veterans Lung Administration Lung Study Group (VALG) staging;
5. At least had progressive disease during or after platinum-based first-line chemotherapy or chemoradiotherapy, and with clear evidence of radiographic progression.

Exclusion Criteria:

1. Previous exposure to immune-mediated therapy; previous use of taxane chemotherapy;
2. Received the last anti-tumor therapy (chemotherapy, radiotherapy) within 4 weeks prior to the first dose of study drug;
3. Received any investigational agent within 4 weeks prior to the first dose of study drug;
4. Received systemic treatment with Chinese herbal medicine indicated for cancer or drugs used for immunoregulation (including thymosin, interferon, interleukin, except for local use for pleural effusion) within 2 weeks before the first dose;
5. Are participating in another interventional clinical study, or observational (non-interventional) clinical study or in the follow-up phase of an interventional study;
6. Pregnant or breastfeeding woman.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Adverse events | 3 months
  The incidence rate of all treatment-emergent adverse events (TEAEs), immune-related adverse events (irAEs) and serious adverse events (SAEs), treatment-related adverse events (TRAEs) and the severity.
Objective remission rate | 12 months
  Proportion of subjects with complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Continuous remission time (DOR) | 12 months
  For subjects with CR or PR, it is defined as the time from the first documented objective tumor response (CR or PR) to objective disease progression (PD) or death.
Disease Control Rate (DCR) | 12 months
  Proportion of subjects with complete response (CR), partial response (PR), or stable disease (SD).
Time to response (TTR) | 12 months
  Time from randomization to first objective tumor response (CR or PR).
Progression-free survival (PFS) | 12 months
  Defined as the time from randomization to the first occurrence of objective disease progression or death.
Overall survival (OS) | 12 months
  Defined as the time from randomization to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cheng, Ph.D, Principal Investigator — Jilin Povince Cancer Hospital
Locations (1):
- Jilin Povince Cancer Hospital, Changchun, Jilin, China